CLINICAL TRIAL: NCT02875080
Title: A Single-center, Open-label, Randomized, Three-way, Crossover Trial to Evaluate the Bioavailability of Brexpiprazole (OPC-34712) Orally Disintegrating Tablets Relative to Brexpiprazole (OPC-34712) Conventional Tablets in Healthy Male Subjects
Brief Title: Evaluation Study of the Bioavailability of Brexpiprazole Orally Disintegrating Tablets in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 331-102-00019; JapicCTI-163351 (Other: Japic)
Record Dates: First submitted 2016-08-08; First posted 2016-08-23 (Estimated); Results first posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Healthy Adult Male
MeSH Terms: interventions — brexpiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- OPC-34712 disintegrating tablet with water (Experimental): OPC-34712 (4 mg) orally disintegrating tablet is administered with water.
  Interventions: Drug: OPC-34712
- OPC-34712 disintegrating tablet without water (Experimental): OPC-34712 (4 mg) orally disintegrating tablet is administered without water.
  Interventions: Drug: OPC-34712
- OPC-34712 conventional tablet with water (Experimental): OPC-34712 (4 mg) conventional tablet is administered with water.
  Interventions: Drug: OPC-34712

INTERVENTIONS:
Drug: OPC-34712
  Other Names: Brexpiprazole

SUMMARY:
The ratios of the geometric means of the ODT formulation to those of the reference formulation (conventional tablet) for the bioavailability variables (Cmax, AUCt, and AUC∞ of brexpiprazole (OPC-34712)).

ELIGIBILITY:
Inclusion Criteria:

* Capable of providing written informed consent prior to initiation of any trial-related procedures, and able, in the opinion of the investigator, to comply with all requirements of the trial

Exclusion Criteria:

* Clinically significant abnormality at the time of screening (eg, significant deviation from reference ranges) or in medical history that, in the opinion of investigator or sponsor may place the subject at risk or interfere with outcome variables, including drug absorption, distribution, metabolism, and excretion
* History of serious mental disorder
* History of drug or alcohol abuse within 2 years prior to screening
* History of any significant drug allergy
* Use of an investigational drug within 120 days prior to the first dosing of trial drug
* Use of tobacco products or daily exposure to secondhand smoke within 2 months prior to screening
* Consumption of grapefruit, grapefruit products, Seville oranges, Seville orange products, starfruit, or starfruit products within 72 hours prior to dosing
* Use of prescription, over-the-counter, or herbal medication, vitamin supplements, or St. John's Wort within 14 days prior to the first dosing of trial drug, or of antibiotics within 30 days prior to the first dosing of trial drug
* History of major surgery of the digestive tract (excluding appendectomy)
* Any subject who, in the opinion of the investigator, should not participate in the trial

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-09-27 (Actual); Primary Completion 2016-11-27 (Actual); Study Completion 2016-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiroaki Ono, Mr, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Kyusyu Region, Japan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 33 subjects were screened for participation in this trial. Of the 33 subjects, 18 subjects were enrolled and randomized to one of 3 sequences, each consisting of 6 subjects. Of the 6 subjects in the Sequence 1 group, 6 subjects received a single dose of OPC-34712 orally disintegrating tablet (ODT) without water, 5 subjects received a single dose of OPC-34712 conventional tablet, and 4 subjects received a single dose of OPC-34712 ODT with water.
Groups:
- Sequence 1: Subjects randomized to Sequence 1 received an ODT without water on Day 1, a conventional tablet on Day 21, and an ODT with water on Day 41.
- Sequence 2: Subjects randomized to Sequence 2 received an ODT with water on Day 1, an ODT without water on Day 21, and a conventional tablet on Day 41.
- Sequence 3: Subjects randomized to Sequence 3 received a conventional tablet on Day 1, an ODT with water on Day 21, and an ODT without water on Day 41.
Period: Overall Study
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Started | 6 | 6 | 6
Completed | 4 | 6 | 6
Not Completed | 2 | 0 | 0
Not completed — Positive urine test for cotinine on Day 20 or Day 40 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (5.5) | 29.7 (7.4) | 28.7 (8.0) | 30.4 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 6 | 6 | 6 | 18
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 6 | 6 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of OPC-34712
Description: To evaluate Cmax of OPC-34712 4-mg ODT formulation relative to 4-mg conventional tablet formulation
Time Frame: Predose, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 48, 72, 96, 120，144, 168, 216, 264, and 312 hours postdose
Population: Pharmacokinetic analysis set consisted of subjects with all evaluable PK parameters from enrolled subjects who had evaluable plasma concentrations. No data imputation was done for missing data, ie, missing data remained missing for the analyses.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OPC-34712 Disintegrating Tablet With Water | OPC-34712 Disintegrating Tablet Without Water | OPC-34712 Conventional Tablet With Water
Number analyzed (Participants) | 15 | 17 | 17
ng/mL | 47.4 (10.0) | 44.9 (13.8) | 46.1 (10.8)

2. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUC∞) of OPC-34712
Description: To evaluate AUC∞ of OPC-34712 4-mg ODT formulation relative to 4-mg conventional tablet formulation
Time Frame: Predose, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 48, 72, 96, 120，144, 168, 216, 264, and 312 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng·h/mL
Arm/Group | OPC-34712 Disintegrating Tablet With Water | OPC-34712 Disintegrating Tablet Without Water | OPC-34712 Conventional Tablet With Water
Number analyzed (Participants) | 15 | 17 | 17
ng·h/mL | 2920 (1630) | 2830 (1270) | 2770 (1460)

ADVERSE EVENTS:
Time Frame: From the start of IMP administration throughout follow-up period (up to 22 days after the last dose of IMP)
Description: A treatment-emergent adverse event (AE) was defined as an AE that started after start of IMP, or an AE that continued from baseline and became serious, IMP-related, or resulted in death, discontinuation, interruption or reduction of trial medication. The safety analysis dataset included all subjects that were administered at least one dose of IMP.
Arm/Group | OPC-34712 Disintegrating Tablet With Water | OPC-34712 Disintegrating Tablet Without Water | OPC-34712 Conventional Tablet With Water
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 8/16 | 7/18 | 9/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-34712 Disintegrating Tablet With Water (N=16) | OPC-34712 Disintegrating Tablet Without Water (N=18) | OPC-34712 Conventional Tablet With Water (N=17)
Nausea (Gastrointestinal disorders) | 4 | 5 | 4
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Orthostatic Hypotension (Vascular disorders) | 4 | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No